CLINICAL TRIAL: NCT06037239
Title: Phase I/II Study of Linperlisib in Combination With Chidamide for Relapsed and Refractory Cutaneous T-cell Lymphoma: a Prospective, Single-center Study
Brief Title: Phase I/II Study of Linperlisib Plus Chidamide for R/R Cutaneous T-cell Lymphoma: a Prospective, Single-center Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-015
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-07

CONDITIONS: Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linperlisib + Chidamide (Experimental): Linperlisib combined with chidamide
  Interventions: Drug: Linperlisib in combined with Chidamide

INTERVENTIONS:
Drug: Linperlisib in combined with Chidamide — Phase 1: dose escalation phase. Drug Linperlisib: 3 dose level of 40mg, 60mg, 80mg qd; Drug Chidamide: fixed dose of 20mg twice weekly.
  Phase 2：dose expansion phase. Drug Linperlisib: RP2D established in the phase I study; Drug Chidamide: fixed dose of 20mg twice weekly in a 4-week cycle

SUMMARY:
HDAC inhibitor chidamide and PI3K inhibitor linperlisib has shown clinical activity as mono therapy in PTCL. The combination of duvelisib and romidepsin is highly active against relapsed and refractory T-cell lymphomas including cutaneous T-cell lymphomas (CTCLs). The aim of this study is to further explore the efficacy and safety of HDAC inhibitor chidamide combined with PI3K inhibitor linperlisib in the treatment of relapsed and refractory CTCLs.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75;
* Mycosis fungoides and Sezary syndrome confirmed by histopathology;
* Patients with measurable lesions, with or without extra-cutaneous lesions, and clinical stage IIB-IVB;
* No remission or relapse after at least one systemic therapy (including total body electron irradiation, becarodine, retinoic acid, interferon, photoseparation and replacement, methotrexate, chidamide, etc.);
* ECOG score of 0-2;
* Adequate bone marrow hematopoietic function: neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥80×109/L, hemoglobin (HGB) ≥90g/L;
* Adequate organ function: NYHA grade 1-2, LVEF≥50%, ALT<2.5UNL, TBil<1.5ULN, SPO2 > 93%@RA, SCr>60ml/(min·1.73m2);

Exclusion Criteria:

* Acute myocardial infarction or unstable angina, congestive heart failure, symptomatic arrhythmia, and significantly prolonged QT interval (> 450ms in men and > 470ms in women) within 6 months;
* Uncontrolled active infections;
* Active hepatitis B and C infection (hepatitis B virus DNA over 1×103 copies /mL is excluded, hepatitis C virus RNA over 1×103 copies /mL is excluded)
* Pregnant or lactating women;
* Investigators judged that they were not suitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D)（Phase 1） | 4 weeks since the date of first dose
  Recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) will be established according to the incidence of dose-limiting toxicities (DLTs) of escalated doses of linperlisib.
Objective response rate (ORR)（Phase 2） | evaluated every 3 months (up to 24 months）

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off (up to 5 years)
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to 5 years)
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
complete remission (CR) rate | evaluated every 3 months (up to 24 months）
  Treatment responses were assessed according to the 2014 Lugano classification criteria
adverse events | evaluated every treatment cycle (up to 24 months）
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pang Z, Wang Y, Liu Z, Zhang S, Wei C, Xu Z, Wang Z, Chen H, Liu J, Zhang W. Linperlisib Plus Chidamide in Relapsed or Refractory Cutaneous T-Cell Lymphoma: A Nonrandomized Clinical Trial. JAMA Dermatol. 2025 Sep 1;161(9):923-930. doi: 10.1001/jamadermatol.2025.1926. PMID 40601335